CLINICAL TRIAL: NCT04306146
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Effects on Neurophysiological Biomarkers of CAD-9303 Oral Treatment in Subjects With Schizophrenia and Normal Healthy Volunteers
Brief Title: Study of CAD-9303 in Subjects With Schizophrenia
Acronym: Affinity-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cadent Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAD9303-101
Record Dates: First submitted 2020-03-10; First posted 2020-03-12 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CAD-9303 (Experimental): Capsules of CAD-9303 will be administered as a single or multiple dose(s). The initial dose will be 3 mg up to 1000 mg total daily dose.
  Interventions: Drug: CAD-9303
- Placebo (Placebo Comparator): Matching placebo will be provided in capsules and administered as a single or multiple dose(s).
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: CAD-9303 — Capsules filled with CAD-9303 from 3 mg up to 1000 mg.
  Arms: CAD-9303
Drug: Placebos — Capsules
  Arms: Placebo

SUMMARY:
This study will consist of Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) cohorts that will be randomized, double-blind, and placebo-controlled to assess the safety, tolerability, and pharmacokinetics of CAD-9303. The first SAD cohort will be in healthy volunteer subjects. The remaining cohorts will be in participants with schizophrenia.

DETAILED DESCRIPTION:
This study will be conducted in two Parts. Part 1 will consist of Single Ascending Dose (SAD) cohorts that will be randomized, double-blind, and placebo-controlled to assess the safety, tolerability, and pharmacokinetics of CAD-9303. Part 2 will consist of Multiple Ascending Dose (MAD) cohorts that will be randomized, double blind, and placebo-controlled to assess the safety, tolerability, and pharmacokinetics of CAD-9303. The effects of CAD-9303 will be explored on event-related potential (ERP), and on sensory and cognitive function. The first SAD cohort will be in healthy volunteer subjects. The remaining cohorts will be in participants with schizophrenia. Participants will meet specified eligibility criteria.

SAD Cohorts will be comprised of 8 subjects; 6 subjects will be administered CAD-9303, and 2 subjects will be administered matching placebo. MAD Cohorts will be comprised of 12 subjects; 9 subjects will be administered CAD-9303, and 3 subjects will be administered matching placebo.

Potential subjects will undergo a screening period (up to 28 days), baseline assessments on Day -3, -2 and -1, and dosing on Day 1 for SAD and Days 1 - 14 for MAD. A follow-up visit will occur 7 days after the last dose. The total duration of individual subject participation may be up to 5 weeks for SAD and 7 weeks for MAD, depending on the duration of the screening period.

The study will assess safety by adverse events, vital signs, laboratory parameters (including chemistry, hematology and urinalysis) and electroencephalogram (EEG); pharmacokinetics of CAD-9303; and exploratory efficacy measures effects on neurophysiological biomarkers, cognitive and negative symptoms.

ELIGIBILITY:
Key Inclusion Criteria:

* For SAD Cohorts: able to tolerate washout from antipsychotic medications for the duration of the planned cohort.
* For MAD Cohorts: not taking an antipsychotic medication at screening and throughout participation in the study or taking one antipsychotic medication at least 6 weeks prior to screening and as a concomitant antipsychotic medication throughout participation in the study.
* Diagnosis of schizophrenia by Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria with duration of illness > 1 year since diagnosis.
* Clinical history of minimal, stable positive symptoms while under treatment with a stable psychotropic regimen.

Key Exclusion Criteria:

* Abnormal findings on screening safety EEG or lifetime history of seizures or stroke.
* Meets current criteria of any psychiatric diagnosis other than schizophrenia, or lifetime history of any psychiatric diagnosis other than schizophrenia based upon the Mini International Neuropsychiatric Interview (MINI).
* Participants with moderate to severe extrapyramidal symptoms including tardive dyskinesia (Simpson-Angus Scale>6, any Abnormal Involuntary Movement Scale (AIMS) Item 1-7 >2), and akathisia (Barnes Akathisia Rating Scale [BARS] Item 4 ≥1).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Assess safety and tolerability of CAD-9303 in participants with schizophrenia and normal healthy volunteers (NHV) | Day 1 through Day 7 Follow-up
  Incidence of Adverse Events

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Collaborative Neuroscience Research, Long Beach, California
  - Hassman Research Institute, Marlton, New Jersey

IPD SHARING:
Plan to Share IPD: No